CLINICAL TRIAL: NCT04091464
Title: TRAIN-BW: Backward Walking Training in Multiple Sclerosis
Acronym: TRAIN-BW
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Nora Fritz, Associate Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URG20192020
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic; Accidental Fall
Keywords: Backward Walking; Neurorehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAIN-BW (Experimental): 1x/week for 8 weeks + home exercise program
  Interventions: Behavioral: Backward Walking Training
- TRAIN-FW (Active Comparator): 1x/week for 8 weeks + home exercise program
  Interventions: Behavioral: Forward Walking Training

INTERVENTIONS:
Behavioral: Backward Walking Training — Training will consist of BW training on both a treadmill and overground. All participants will receive 1x/week training with a trained member of the research team, who will progress the participant week-to-week and ensure safety. Treadmill speed will be determined by baseline BW walking speed and incrementally increased with each training week to subject tolerance. Participants will follow a home exercise program for the remainder of the week that includes BW, backward stepping, and functional exercises that incorporate BW movements.
  Arms: TRAIN-BW
Behavioral: Forward Walking Training — Training will consist of FW training on both treadmill and overground. All participants will receive 1x/week training with a trained member of the research team, who will progress the participant week-to-week and ensure safety. Treadmill speed will be determined by baseline FW walking speed and incrementally increased with each training week to subject tolerance. Participants will follow a home exercise program for the remainder of the week that includes FW, forward stepping, and functional exercises that incorporate FW movements.
  Arms: TRAIN-FW

SUMMARY:
Individuals with multiple sclerosis (MS) experience in impairments in mobility and cognition that increase the risk for accidental falls. More than 50% of individuals with MS experience injurious falls within a 6-month period. Current interventions to improve fall risk have focused on forward walking (FW) and balance training, resulting in small declines in the relative risk for falls with a large degree of variability. Interestingly, motor differences between MS and healthy controls are more pronounced in backward walking (BW), yet no studies have investigated BW training as an intervention to reduce fall risk in persons with MS. This study will investigate the feasibility, acceptability and impact of BW training compared to forward walking training on motor function and fall risk in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS
* PDDS <6, indicating ability to ambulate with or without an assistive device >/= 50% of the time
* Self-reported walking dysfunction as evidenced by a score of >/= 30 on MSWS-12 OR reports of 2 or more falls in the prior 6 months, indicating a frequent faller.

Exclusion Criteria:

* MS relapse within the past 30 days
* comorbid neurological disorder
* acute orthopedic disorder/injury
* unable to follow study-related commands

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Sway during quiet stance | Change in sway at 8 weeks
  Measured with APDM Sensors
Stepping latency on push-and-release test | Change in stepping latency at 8 weeks
  Measured with APDM Sensors

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | 8 weeks
  Scores range from 8-32, with high scores indicating greater satisfaction with the intervention
Patient Global Impression of Change | 8 weeks
  Perceived Treatment Effect; scores range from 1-7 with higher scores indicating greater perception of improvement related to the intervention.
Number of Active Minutes | Change in Physical Activity measures at 8 weeks
  Measured with Accelerometry, passively collected for a 1 week period prior to the intervention and again after the intervention concludes 8 weeks later.
Number of Falls | 6 months
  Number of falls reported in 6 month period after the intervention ends
Forward and Backward Velocity and Double Support Time | Change in velocity and double support time at 8 weeks
  Walking speed and double support time (spatiotemporal measures of gait)
ABC Scale | Change in balance confidence at 8 weeks
  Balance confidence

CONTACTS AND LOCATIONS:
Overall Officials: Nora Fritz, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No